CLINICAL TRIAL: NCT01278602
Title: A Multi-center Phase II Study of R-ESHAP Followed by Autologous Transplantation as Salvage Treatment for Patients With Refractory or Relapsed Diffuse Large B-cell Lymphoma.
Brief Title: R-ESHAP Followed by Autologous Transplantation for Refractory or Relapsed Diffused Large B-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ye Guo, Dr., Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LMTG 11-01
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Diffuse large B-cell lymphoma; Chemotherapy; R-ESHAP; Autologous stem cell transplantation
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- R-ESHAP (Experimental): Rituximab 375mg/m2 at day 0, Meththylprednisolone 500mg IV at days 1 to 5, Etoposide 40mg/m2 at days 1 to 4, Cisplatin 25mg/m2 at days 1 to 4, Cytarabine 2000mg/m2 at day 5. Frequence of cycles: every 3 weeks. Numbers of cycles: 3 cycles.
  Interventions: Drug: R-ESHAP

INTERVENTIONS:
Drug: R-ESHAP — Rituximab 375mg/m2 at day 0, Meththylprednisolone 500mg IV at days 1 to 5, Etoposide 40mg/m2 at days 1 to 4, Cisplatin 25mg/m2 at days 1 to 4, Cytarabine 2000mg/m2 at day 5. Frequence of cycles: every 3 weeks. Numbers of cycles: 3 cycles.
  Other Names: Mabthera

SUMMARY:
The aim of study is to prove R-ESHAP regimen followed by autologous stem cell transplantation as salvage treatment in patients with refractory or relapsed diffuse large B-cell lymphoma is effective.

DETAILED DESCRIPTION:
The standard treatment in patients with refractory or relapsed diffuse large B-cell lymphoma is salvage chemotherapy followed by autologous transplantation for responsive patients. However, the standard of salvage chemotherapy remains uncertain. This study is to evaluate the efficacy and safety of R-ESHAP regimen in a multi-center basis.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18-65 years old
* Histological confirmed diffuse large B-cell lymphoma
* Refractory or first relapsed disease
* Prior anthracycline exposure
* Measurable disease
* ECOG performance status 0-1
* Life expectancy of more than 3 months
* Bone marrow function: ANC≧1.5×109/L, PLT≧100×109/L, Hb≧90g/L
* Liver function: total bilirubin, ALT and AST <1.5×UNL
* Renal function: Cr<1.5×UNL, CCR≧50ml/min
* No contraindication for transplantation

Exclusion Criteria:

* Evidence of CNS and bone marrow involvement
* More than 1 type of chemotherapy regimens exposure
* High level of HBV DNA
* Contraindication of high-dose methylprednisolone
* Pregnant or lactating women
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* History of allergic reaction/hypersensitivity to rituximab
* Significant active infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 6 weeks

SECONDARY OUTCOMES:
3-year progression-free survival rate | 3 years
3-y overall survival rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China